CLINICAL TRIAL: NCT06091826
Title: Phase II Study Assessing Efficacy and Safety of NFL-101 on Reduction of Reinforcing Properties of Cigarettes (PRECESTO Trial)
Brief Title: Study Assessing Efficacy and Safety of NFL-101 on Reduction of Reinforcing Properties of Cigarettes (PRECESTO)
Acronym: PRECESTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NFL Biosciences SAS (Industry)
Responsible Party: Principal Investigator, Yves Donazzolo, MD Eurofins Optimed, NFL Biosciences SAS
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: v1.2
Record Dates: First submitted 2023-02-21; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Tobacco Products; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NFL-101 (Experimental): 100 μg per subcutaneous injection (in each arm), two injections at day 1
  Interventions: Drug: NFL-101
- Placebo (Placebo Comparator): Water for Injection (WFI), two injections at day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NFL-101 — Subcutaneous injections
  Other Names: Tobacco leaf extract
  Arms: NFL-101
Drug: Placebo — Subcutaneous injections
  Other Names: Water for injection
  Arms: Placebo

SUMMARY:
PRECESTO is a randomized, double-blind, cross-over trial on 34 smokers who do not want to stop smoking and get high satisfaction from smoking.

The primary objective is to assess efficacy of NFL-101 in reducing the positive reinforcing properties of cigarettes compared to placebo measured by the modified Cigarette Evaluation Questionnaire (mCEQ) "Smoking Satisfaction" (items 1, 2, and 12) subscale.

DETAILED DESCRIPTION:
PRECESTO is a monocentric, placebo-controlled, randomized and double-blind Phase 2a exploratory study, with a crossover covering two periods of 28 days each, including 34 smokers who do not want to quit and have high smoking satisfaction. Each participant is his or her own control and receives, on a random and alternating basis, either NFL-101 or the placebo at the start of each of the two periods. At the end of the study, all the participants received one dose of NFL-101 and one dose of the placebo. For each participant, the order in which NFL-101 and the placebo are administered is kept secret. For each period, the participants receive the treatments on day 1 (D1) then answer, with complete independence, the modified Cigarette Evaluation Questionnaire (mCEQ) on days 4 (D4), 7 (D7), 14 (D14), 21 (D21) and 28 (D28).

The objective is to assess the safety and efficacy of NFL-101 as a pretreatment for smoking cessation, NFL-101 beeing administered a few days or weeks before a quit attempt while smokers are asked to smoke ad libitum (meaning to continue either to try to smoke the same amount or to smoke freely). It is indeed recognized that reducing satisfaction from smoking before a quit attempt begins to undermine the learned association between smoking and reward and thus promotes the success of these attempts.

ELIGIBILITY:
Inclusion Criteria:

* Equipped with a web connection via a computer or tablet;
* Subject currently smoking at least 10 cigarettes per day;
* Exhaled CO ≥ 9 ppm;
* Subject with a mCEQ Satisfaction subscale score ≥ 4
* Subject not wanting to stop smoking (MTSS score ≤ 2)
* Subject not under tobacco cessation therapy since at least 30 days;
* Considered as healthy for the study after a comprehensive clinical assessment (detailed medical history and complete physical examination);
* For women of childbearing potential: commitment to consistently and correctly use of a highly effective contraceptive measure: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner or sexual abstinence for the duration of the trial;
* Females of non-childbearing potential: either surgically sterilized or at least 1 year postmenopausal (amenorrhea duration at least 12 months);
* Negative pregnancy test at screening visit;
* Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests). Individual values out of the normal range can be accepted if judged clinically non relevant by the investigator;
* Negative prick test at screening visit for the whole study product (extract of Tobacco leaf and NaCL), and positive for histamine;
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research;
* Subject having signed the informed consent agreement.

Exclusion Criteria:

* Pregnancy and breastfeeding;
* Concomitant participation to another clinical trial;
* Concomitant active infectious diseases;
* Suicidal or depressive state
* Positive results of screening for drugs of abuse
* History or presence of drug or alcohol abuse (alcohol consumption > 40 grams / day);
* Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study (for subjects in France only);
* Subject who, in the judgment of the investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change of smoking satisfaction | at Day 4
  Success in achieving a 1 point reduction in the mCEQ "Smoking Satisfaction" subscale

SECONDARY OUTCOMES:
Change of smoking satisfaction | at Day 7, at Day 14, at Day 21 and at Day 28
  Success in achieving a 1 point reduction in mCEQ "Smoking Satisfaction" subscale
Change in psychological reward, aversion, enjoyment of respiratory tract sensation and craving | at Day 4, at Day 7, at Day 14, at Day 21 and at Day 28
  Success in achieving a 1 point reduction in mCEQ "Psychological Reward"; "Aversion"; "Enjoyment of Respiratory Tract Sensations"; and "Craving Reduction" subcales
"Have you found your urges to smoke stronger or weaker than usual in the last 24 hours?" | at Day 4, at Day 7, at Day 14, at Day 21 and at Day 28
  With response options of "much stronger," "slightly stronger," "same as before," "slightly weaker," and "much weaker"
"Have you found cigarettes more or less enjoyable than usual in the last 24 hours?" | at Day 4, at Day 7, at Day 14, at Day 21 and at Day 28
  With response options of "much more enjoyable," "slightly more enjoyable," "same as before," "slightly less enjoyable," and "much less enjoyable"
Preference question : "Is there one of the two administrations that made you want to quit smoking or reduce your cigarette consumption more than the other?" | at EOS visit
  With response options of administration 1, administration 2, I dont know, imponderable factors (for example covid, death of a relative, job loss, etc.) do not allow me to answer

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, Isère, France

IPD SHARING:
Plan to Share IPD: No